CLINICAL TRIAL: NCT05972187
Title: The Effect of the Indoor Environmental Quality (IEQ) on Cognition and Health
Brief Title: The Effect of IEQ on Cognition and Health
Acronym: IEQ-HUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL81104.068.22
Record Dates: First submitted 2023-03-24; First posted 2023-08-02 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2023-09

CONDITIONS: Environmental Exposure; Temperature Change, Body; Condition; Healthy
Keywords: Temperature; Humidity; Thermoregulation; Cognition; Health
MeSH Terms: conditions — Body Temperature Changes; Disease | interventions — Temperature; Humidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Temperature and Humidity (Experimental): 32C or 25C and 30%RH or 70%RH
  Interventions: Other: Temperature and Humidity

INTERVENTIONS:
Other: Temperature and Humidity — Temperature and Humidity of room changed

SUMMARY:
The goal of this study is to learn about the effect of heat and humidity on cognition and health. The main question[s] it aims to answer are:

type of study: interventional participant population: 20-40years, both gender, healthy Participants will be exposed for 4 different sessions of 8 hours at a time, to 32˚ C or 25˚ C in combination with relative humidity of 30 %RH or 70 %RH.

DETAILED DESCRIPTION:
Overall, the project aims to evaluate the effects of high vs. neutral temperature (32˚ C vs. 25˚ C) in combination with high vs. low humidity (30 %RH vs. 70 %RH) on cognition, for longer exposure duration (8 hours). Deviations from the personal comfort zones are expected to affect both subjective feelings and physiological parameters. Therefore, the following parameters will be included: cognition, environmental perception, energy expenditure, body temperatures.

Main research question and primary objective:

What is the impact of being exposed for 8 hours to a high humidity (RH 70%) versus low humidity (RH 30%) on cognitive performance of individuals if the room temperature is 25ºC or 32ºC?

This leads to the following hypotheses:

* Exposure to an indoor high relative humidity (RH 70%) at a warm temperature (32ºC) of a long duration (8 hours) reduces the composite score, speed and accuracy of cognitive performance compared to an exposure to a low RH (30%) at the same temperature (32ºC) due to the humidity.
* An exposure to an indoor high relative humidity (RH 70%) at a neutral temperature (25ºC) of a long duration (8 hours) would reduce the composite score, speed and accuracy of cognitive performance compared to an exposure to a low RH (30%) at a neutral temperature (25 ºC) due to previous literature for humidity influences at neutral temperatures.

Secondary research question and secondary objective:

What is the effect of high vs. neutral temperature (32˚ C vs. 25˚ C) in combination with high vs. low humidity (30 %RH vs. 70 %RH) on physiological responses, environmental perception, decision making, and bias behaviour?

This leads to the following hypotheses:

1. Does an 8 hour exposure to an elevated concentration of indoor humidity lead to an increase in energy expenditure and/or a greater difference in proximal and distal blood flow and skin temperature gradients compared to a lower indoor humidity for each of the temperature settings?
2. What are the effects of high humidity on substrate oxidation, blood pressure, heart rate variability, proximal and distal skin temperature, risk behavior and decision-making responses of individuals?
3. What are the effects of higher humidity on environmental perception (thermal, air quality, moisture/wetness) comfort, perception, and sensation?

   * An exposure to an indoor high relative humidity (RH 70%) at a warm temperature (32ºC) of a long duration (8 hours) reduces the composite score, speed and accuracy of cognitive performance compared to an exposure to a high RH (70%) at a neutral temperature (25 ºC) due to the humidity and temperature.
   * An exposure to an indoor low relative humidity (RH 30%) at a warm temperature (32ºC) of a long duration (8 hours) would reduce the composite score, speed and accuracy of cognitive performance compared to an exposure to the same low RH (30%) at a neutral temperature (25 ºC) due to the temperature.

Exploratory research question and objective:

What is the interaction effect of high vs. neutral temperature (32˚ C vs. 25˚ C) in combination with high vs. low humidity (30 %RH vs. 70 %RH) on cognitive performance, physiological responses, environmental perception, decision making, and bias behaviour?

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5-26 kg/m2
* Age between 20-40 years
* Proficient with the English language in both verbal and written form
* Healthy; no illness or disease or prescribed medication within the last 3 months
* Steady dietary and sleeping habits
* Regularly physically active (i.e., regularly active but less than 3 times a week for less than 2 hours per session at moderate intensity)
* Non-smoker or person who quit smoking more than five years ago
* Reside in the Netherlands (or surrounding countries) for at least 6 months

Exclusion Criteria:

* Subjects with cardiac problems and cardiovascular diseases, such as angina pectoris, cardiac infarction, and arrhythmias
* Subjects with any medical condition requiring treatment and/or medication (except oral contraceptives) that might interfere with the investigated parameters E.g., Extreme chronotype, colour blindness, epilepsy
* Subjects with a disorder or disease (Parkinson, Attention Deficit Hyperactivity Disorder (ADHD), Alzheimer, diabetes, cardiovascular disorder, respiratory impairments (for example asthma), hypertension, obesity, or any other condition that can impair the lung function), or Raynaud's phenomenon
* Subjects with abnormal diet and sleeping patters and/or abnormal body weight (weight gain or loss >3kg in the past month)
* Subjects who recently participated in other interventional biomedical study within 1 month prior to screening visit
* Subjects, who do not want to be informed about unexpected medical findings, or do not wish that their treating physician will be informed, cannot participate in this study
* Subjects with previous covid infection in the past 3 months or any subject with persistent long covid symptoms that may have caused ongoing loss of or altered sense of smell
* Subjects who had severely altered sleep patterns in the past year
* Subjects employed with night shift work within the past year
* Subjects who consume more than two standard drinks of alcohol per day
* Subjects who consume more than two standard drinks of coffee per day
* Subjects who are pregnant

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-06-18 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Cognition | 1 month
  Using a tablet based cognitive test battery

SECONDARY OUTCOMES:
Heart Rate (bpm) | 1 month
  Heart Rate measured using Polar heart rate belt in (bpm) with RR and ECG data extracted
Blood pressure (mmHg) | 1 month
  Blood pressure - both systolic and diastolic pressures measured hourly using an automated blood pressure monitor and cuff
Metabolic Rate (ml O2//min/kg) | 1 month
  Metabolic rates measured through whole room calorimetry
Skin Temperature (C) | 1 month
  Skin temperature measured using thermochron (ibuttons) at multiple sites
Body Core Temperature (C) | 1 month
  Core Temperature measured via telemetric pill ingested in the morning

OTHER OUTCOMES:
Room Temperature (C) | 1 month
  Environmental measures are measured continuously using temperature specific sensors in the room
Humidity (%) | 1 month
  Environmental measures are measured continuously using humidity specific sensors in the room

CONTACTS AND LOCATIONS:
Overall Officials: Guy Plasqui, PHD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
If requested raw data will be provided.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Ongoing, depends on the request.
Access Criteria: Official request made stating the purpose of use for the data. Only individuals that consent to their data to be used in further analysis will be shared.